CLINICAL TRIAL: NCT03245320
Title: A Post-Market Observational Study to Evaluate Performance and Safety of the TITAN™ Total Shoulder System
Brief Title: Clinical Evaluation of the TITAN™ Total Shoulder System
Status: Terminated | Type: Observational
Why Stopped: Terminated by the Sponsor. Decision not due to adverse events, complications, or device issues.
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: T-TSS-002
Record Dates: First submitted 2017-05-03; First posted 2017-08-10 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Arthritis; Arthritis, Degenerative; Rheumatoid Arthritis; Post-traumatic Arthrosis of Other Joints, Shoulder Region; Rotator Cuff Syndrome of Shoulder and Allied Disorders; Fracture; Avascular Necrosis; Joint Instability; Joint Trauma; Dislocation, Shoulder; Pain, Shoulder
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Fractures, Bone; Osteonecrosis; Joint Instability; Shoulder Dislocation; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- TITAN™ Total Shoulder System Generation 1.0: Integra TITAN™ Total Shoulder System Generation 1.0
  Interventions: Device: Integra TITAN™ Total Shoulder Generation 1.0

INTERVENTIONS:
Device: Integra TITAN™ Total Shoulder Generation 1.0 — Total Shoulder Arthroplasty or Hemiarthroplasty

SUMMARY:
A post market, non-randomized, multi-center, open-label,clinical study using survivorship to study the safety and efficacy of the Integra® TITAN™ Total Shoulder System 1.0 (TAS) when used for total shoulder arthroplasty.

DETAILED DESCRIPTION:
Observational, multi-center, post-market study to provide data on the performance and safety of the TITAN™ Total Shoulder System. The study will enroll patients that underwent total shoulder arthroplasty with the TITAN™ Total Shoulder System per standard of care less than 5 years ago. Available retrospective data up to the 2-year time point will be collected, per the study protocol, from medical record reviews. Prospective observational data will be collected from the time of patient enrollment during the following postoperative clinical visits: 1 year, 2 years, 5 years and 10 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has undergone shoulder arthroplasty with the first generation TITAN Total Shoulder System.
2. The first generation TITAN Total Shoulder System is still intact and the subject has not received any revision surgeries involving the TITAN Total Shoulder System.
3. Subject is willing and able to participate in required follow-up visits at the investigational site and to complete study procedures.

Exclusion Criteria:

1. Subject, in the opinion of the PI, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study such as mental illness, or drug or alcohol abuse.
2. Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject has undergone shoulder arthroplasty with the first generation TITAN Total Shoulder System.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Implant survival at 2 years | 2 years
  Implant survivorship is defined as absence of device removal or revision of one or more of the implant component(s).

SECONDARY OUTCOMES:
Implant survival . | 5 and 10 years
  Implant survivorship is defined as absence of device removal or revision of one or more of the implant component(s).
Relative change of Range of Motion (ROM) compared to baseline | 2, 5, and 10 years
  Relative change of Range of Motion (ROM) compared to baseline
Radiographic assessment | 2, 5, and 10 years
  Radiographic assessment for loosening, malpositioned implant, subsidence, subluxation, and radiolucency
Relative change in Quality Of Life (EQ-5D) compared to baseline | 2, 5, and 10 years
  Relative change in Quality Of Life (EQ-5D) compared to baseline
Relative change of American Shoulder and Elbow Surgeon Score (ASES) compared to baseline | 2, 5, and 10 years
  Relative change of American Shoulder and Elbow Surgeon Score (ASES) compared to baseline
Relative change of PENN Pain and Function Score (PENN) compared to baseline | 2, 5, and 10 years
  Relative change of PENN Pain and Function Score (PENN) compared to baseline
Relative change in Quality Of Life (SF-12V1) compared to baseline | 2, 5, and 10 years
  Relative change in Quality Of Life (SF-12V1) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tummon, Study Director — Integra LifeSciences
Locations (2):
- United States (2):
  - OrthoIndy, Indianapolis, Indiana
  - The Rothman Institute, Philadelphia, Pennsylvania